CLINICAL TRIAL: NCT03717025
Title: A Comparative Study Between Autologous Mini Punch Grafting, Suction Blister Grafting and Non-Cutured Epidermal Cell Suspension on Resistant Sites in Stable Vitiligo
Brief Title: Comparison of Surgical Methods on Resistant Sites in Stable Vitiligo Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Davinder Parsad, PROFESSOR, DEPARTMENT OF DERMATOLOGY, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT/IEC/2017/1251
Record Dates: First submitted 2018-10-16; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Vitiligo
Keywords: ACRAL
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mini Punch Grafting (Active Comparator)
  Interventions: Procedure: MINI PUNCH GRAFTING
- Suction Blister Epidermal Grafting (Active Comparator)
  Interventions: Procedure: SUCTION BLISTER EPIDERMAL GRAFTING
- Non Cultured Epidermal Cell Suspension (Active Comparator)
  Interventions: Procedure: NON CULTURED EPIDERMAL CELL SUSPENSION

INTERVENTIONS:
Procedure: SUCTION BLISTER EPIDERMAL GRAFTING — 1. Preferred donor sites for making blister is lateral aspect of upper thigh. The area is shaved and cleansed with surgical spirit.
  2. Blister formation is induced by using suction apparatus.
  3. Recipient site is surgically prepared by doing dermabrasion.
  4. After formation of blisters, each blister is gently cleansed with normal saline and cut all along its border with curved iris scissors parallel to the skin surface. The roof is everted over the thumb with dermal surface facing upwards and then with the help of blunt end of forceps it is placed on the recipient area.
  5. The graft is firmly pressed with sterile moist gauze to remove any underneath serous collection.
  6. The pressure dressing is done with double layer framycetin tulle, moist gauze and bandage.
  7. Donor area is dressed with dry sterile pads.
  8. The part is immobilized and Antibiotics and Analgesic are given till dressing are removed (after 5-7 days).
  Arms: Suction Blister Epidermal Grafting
Procedure: MINI PUNCH GRAFTING — 1. Recipient area is prepared first after shaving and cleaning with surgical spirit. 2 % lignocaine with or without adrenalin will be infiltrated as local aneasthetic.
  2. The punched out chambers are spaced at a gap of less than 5 mm (preferably 2 - 2.5 mm) from each other.
  3. The donor area is either upper lateral portion of thigh or gluteal region.
  4. Grafts are placed directly from donor to the recipient area. Care is taken, so that graft edges are not folded, the tissue is not crushed or placed upside down.
  5. Hemostasis is achieved by pressing a saline soaked gauze piece over the area.
  6. For the recipient area 3 layers of dressing from inside out are : paraffin embedded non adherent sterile gauze, sterile surgipad, and micropore.
  7. For the donor area only surgipad and micropore are used.
  8. Immobilisation of recipient area is advised along with antibiotics and analgesics till removal of dressing (after 4-7 days).
  Arms: Mini Punch Grafting
Procedure: NON CULTURED EPIDERMAL CELL SUSPENSION — 1. About one-tenth the size of recipient area is selected as the donor site.
  2. Split thickness skin graft is taken under aseptic precautions with the help of a shaving blade held firmly by a straight artery forceps.
  3. The area is dressed with Bactigras gauze.
  4. Split thickness skin specimen is transferred under aseptic conditions to a container with Normal Saline and transferred to laboratory for preparing suspension.
  5. Recipient site is dermabraded under aseptic precautions until tiny pinpoint bleeding spots are seen.
  6. Epidermal cell suspension is carefully transferred to a tuberculin syringe.
  7. With 18 gauge needle attached to this syringe, suspension is spread evenly on dermabraded recipient site.
  8. This is then covered with Collagen dressing, followed by bactigras, guaze and tegaderm dressings from inside to outside.
  9. The patient is observed for 2 hours after performing the procedure and given antibiotics and analgesics for 5-7 days till dressing removal.
  Arms: Non Cultured Epidermal Cell Suspension

SUMMARY:
Comparing the Efficacy of Three Different Surgical Methods on Resistant Sites in Stable Vitiligo.

DETAILED DESCRIPTION:
The treatment of vitiligo includes both medical and surgical modalities, whose goal is to restore melanocytes to the depigmented skin so that the epidermis restores back to normal morphology and functions. Although medical treatment is the main stay of treatment, it is not effective in all and residual lesions need augmented surgical treatment later for further completion of repigmentation.

Now a day surgical modalities have become treatment of choice for stable vitiligo not responding to medical treatment although there are numerous sites which do not respond that well to surgical procedure as well. The investigators ought to compare the efficacy of 3 well established surgical methods i.e. Mini Punch Grafting vs Suction Blister Epidermal Grafting vs Non Cultured Epidermal cell Suspension on stable vitiligo patches localized to acral areas and bony prominences like elbows, knees and ankles. Out of all the vitiligo patches in a given participant, 3 different patches on acral and bony areas will be chosen and participants will be treated with 3 different methods.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with clinical diagnosis of focal, segmental or generalized vitiligo
2. Patients with lesions of size > 1.5cm x 1cm present on acral areas and bony prominences.
3. Vitiligo lesions has been stable for 1 year.
4. Disease not responding to medical treatment, or there are residual patches (after medical therapy) of vitiligo which inturn are located on acral areas and bony prominences.
5. Maximum size of vitiligo patches to be selected for surgery will not be >100cm2.

Exclusion Criteria:

1. Age less than 18 years
2. Pregnancy and lactation
3. Patient with actively spreading vitiligo
4. History of Koebnerisation
5. History of hypertrophic scars or keloidal tendency
6. Bleeding disorders
7. Patients with unrealistic expectation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Repigmentation At Surgery Site | Repigmentation will be assessed at 12 weeks.
  To assess the difference in extent of repigmentation of the surgery site by three different methods at 12 weeks of post treatment follow up in a given patient.
  Repigmentation will be assessed as follows:
  ≤25% Minimal repigmentation 26-50% Mild repigmentation 51-75% Moderate repigmentation 76-90% Marked repigmentation >90% Excellent repigmentation

SECONDARY OUTCOMES:
Color Matching of Repigmented Area | Assessment at 12 weeks.
  Color matching of the repigmented area with the surrounding normal skin will be done in each case as 'somewhat lighter than', 'same as' or 'somewhat darker than' normal skin.
Patient's Quality of Life Post Surgery | Assessment at 12 weeks.
  Patient satisfaction will be assessed using Patient Global Assessment score.
Patient's Quality of Life Post Surgery | Assessment at 12 weeks.
  Quality of life assessement post procedure will be done using Vitiligo specific questionnaire.
PATTERN OF REPIGMENTATION | Assessment at 12 weeks.
  Pattern of repigmentation attained post-procedure will be noted as 'diffuse', 'perifollicular' or 'migrating from the borders'.
ADVERSE EVENTS | Assessment at 4, 8 and 12 weeks.
  Adverse events both at recipient and donor sites.

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided
Overall results of the study will be available to other researchers.